CLINICAL TRIAL: NCT05155826
Title: The Effect of Virtual Reality for Pain Management During Intracervical Balloon Placement for Labor Induction: a Randomized Controlled Trial (VIRTUALMAG)
Brief Title: Effect of Virtual Reality for Pain Management During Intracervical Balloon Placement for Artificial Childbirth Induction
Acronym: VIRTUALMAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21CH027; ANSM (Other: 2021-A01886-35)
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Delivery Problem; Labor Pain
Keywords: labor induction; intra-cervical balloon; pain; virtual reality; Cook®
MeSH Terms: conditions — Dystocia; Labor Pain; Pain

STUDY DESIGN:
Intervention Model Description: This is a prospective monocentric study, randomized in 2 parallel groups, evaluating the effectiveness of the use of a virtual reality headset on the reduction of pain during intra-cervical balloon insertion for induction versus standard care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (control group) (No Intervention): Patient benefit the standard care during the placement of Cook's balloon (standard care).
- standard care and virtual reality (experimental group) (Experimental): Patient benefit the standard care during placement of Cook's balloon (standard care) with the use of a virtual reality.
  Interventions: Device: Virtual Reality Headset

INTERVENTIONS:
Device: Virtual Reality Headset — The patient will benefit from the placement of Cook's balloon (standard care) with the placement of the virtual reality headset on the examination table with the launch of the software before the beginning of the procedure. The virtual reality helmet will be removed at the end of the procedure.
  Other Names: Deepsen® VRx and Shenzhen Huajin® electronics Co
  Arms: standard care and virtual reality (experimental group)

SUMMARY:
The labor induction concerns 22% of births in France. In the event of labor induction, in almost two thirds of cases, a cervical ripening method is used and the use of mechanical methods is observed for 8% of cervical ripening. Intra-cervical balloon placement is generally well tolerated but is frequently associated with pain and acute anxiety. There are few options for pain relief. Virtual reality, a relatively new intervention, has been studied as a distraction technique for pain relief, but never in the context of the induction of childbirth.

DETAILED DESCRIPTION:
It's prospective single-center, randomized, single-blind, prospective study (1:1, 2 group randomization) comparing a group of patients who benefited from the use of the virtual reality headset to a group of patients who received standard care during balloon insertion. Two groups of patients will be formed: a "standard care" group and a "standard care + virtual reality" group.

The study will take place at the Saint-Etienne University Hospital Center in the gynecology-obstetrics department.

The principal objective is to evaluate the effectiveness of the use of a virtual reality helmet on the reduction of pain during the insertion of an intra-cervical balloon for childbirth induction versus the use of standard care.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman presenting to the Gynecology-Obstetrics Department of the Saint-Etienne University Hospital for an induction by Cook's balloon.
* Patients affiliated or entitled to a social security system
* Patients having given their agreement to participate and after signing the consent form

Exclusion Criteria:

* Woman refusing to participate in the study (lack of consent)
* Non French-speaking woman (impossibility of carrying out a good quality interview of the pregnant woman)
* Women suffering from blindness, deafness or epilepsy against the use of the virtual reality helmet.
* Participation in another interventional study.
* Patient under guardianship or curatorship
* Patient subject to a legal protection measure or unable to express their consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
maximum pain felt during balloon placement | Day: 0
  Measurement of the maximum pain experienced during the placement of the intra-cervical balloon using a numerical scale from 0 to 10: 0 = no pain, 10 = maximum pain.

SECONDARY OUTCOMES:
average pain felt during balloon placement | Day: 0
  Average pain felt during balloon placement measured by a numerical scale from 0 to 10. (0 no pain - 10 maximum pain).
Nociception Level Index (NOL™) during balloon placement | Day: 0
  Measured Nociception Level Index (NOL ™) calculated by the PMD200 Pain Monitor™.
  Nociception Level Index is numerical index from 0 to 100. (>25 = pain)
Anxiety felt during balloon placement | Day: 0
  Anxiety felt during balloon placement measured by a numerical scale from 0 to 10 : 0 = no anxiety - 10 = maximum anxiety.
difficulty of balloon placement by the midwife during induction of labor | Day: 0
  Difficulty of balloon placement by the midwife is measured by questionary classified as very easy / easy / ni easy ni difficult / difficult / very difficult
patient's satisfaction with the use of the virtual reality headset. | Day: 0
  patient's satisfaction is evaluated by Likert scale: Completely satisfied/ Satisfied/ Neutral/ Not satisfied/ Not at all satisfied
midwife's satisfaction with the use of the virtual reality headset. | Day: 0
  midwife's satisfaction is evaluated by Likert scale: Completely satisfied/ Satisfied/ Neutral/ Not satisfied/ Not at all satisfied
tolerance of the virtual reality helmet by the patient. | Day: 0
  Tolerance is a composite outcome : nausea (YES/NO), dizziness (YES/NO), premature stopping (YES/NO)

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine RAIA BARJAT, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No